CLINICAL TRIAL: NCT04377958
Title: Development and Validation of a Serum Biomarker for the Diagnostic Work-up of Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Tatjana Decaesteker, Principal Investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s52549
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Asthma; Biomarkers
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthmatics (Other): Asthmatic group from which serum samples will be collected for analysis
  Interventions: Diagnostic Test: Serum biomarker testing

INTERVENTIONS:
Diagnostic Test: Serum biomarker testing — Serum and sputum samples will be collected and biomarkers will be evaluated using ELISA

SUMMARY:
Serum samples of asthmatic patients will be screened for serum biomarkers

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years
* physician-diagnosed asthma

Exclusion Criteria:

* No clear asthma phenotype
* Presence of other pulmonary diseases (Chronic obstructive pulmonary disease, alfa-1-antitrypsine deficiency emphysema, Immunoglobulin E deficiency, allergic bronchopulmonary aspergillosis)
* > 15 pack years
* No sputum available
* Respiratory infection
* Other inflammatory diseases (Rheumatoid Arthritis, Colitis Ulcerosa)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Serum calprotectin | Day 1
  Serum Calprotectin (pg/ml) will be measured in serum samples using a U-plex assay

SECONDARY OUTCOMES:
Sputum calprotectin | Day 1
  Sputum Calprotectin (pg/ml) will be measured in sputum samples using a U-plex assay

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Dupont, Principal Investigator — UZ Leuven

IPD SHARING:
Plan to Share IPD: No